CLINICAL TRIAL: NCT01005056
Title: Drug Use Investigation of MARVELON
Brief Title: Post-marketing, Observational Study to Confirm the Safety and Efficacy of MARVELON (Study P06083)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P06083
Record Dates: First submitted 2009-08-27; First posted 2009-10-30 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Contraception
MeSH Terms: interventions — Ethinyl Estradiol; Desogestrel

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Marvelon®: Single arm study. All participants receive Marvelon® according to the approved dosage and administration method.
  Interventions: Drug: Ethinylestradiol + Desogestrel

INTERVENTIONS:
Drug: Ethinylestradiol + Desogestrel — All participants receive Marvelon® according to the approved dosage and administration method.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Marvelon® in the prevention of pregnancy.

Post-marketing surveys are not considered applicable clinical trials and thus the results of this survey will not be posted at its conclusion. The results will be submitted to public health officials as required by applicable national and international laws.

DETAILED DESCRIPTION:
Women with willingness to prevent pregnancy, who do not meet any of the contraindications, and who will take Marvelon® in compliance with the approved dosage and administration method will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Women with willingness to prevent pregnancy and to take Marvelon® in compliance with the approved dosage and administration method

Exclusion Criteria:

* Women with constitution of hypersensitivity to ingredients of this product.
* Woman with estrogen-dependent tumor (for instance, breast cancer, cancer of uterine body and uterine myoma), cancer of uterine cervix, or suspected of them. [aggravation or manifestation of tumor may be induced.]
* Patients with abnormal genital bleeding for which diagnosis has not been established [Genital cancer is suspected. If bleeding is due to genital cancer, aggravation or manifestation of cancer may be induced.]
* Patients with thrombophlebitis, embolism pulmonary, cerebrovascular disorder, coronary diseases, or a history thereof [blood coagulation capacity may be increased and these symptoms may be aggravated.]
* Smoker aged 35 years or older taking 15 or more pieces of tobacco per day [It has been reported that cardiovascular disorder including myocardial infarction is liable to occur.]
* Patients with migraine accompanied by signal symptom (scotoma scintillans, star-shaped flash, etc.) [It has been reported that compared with patients without concomitant symptom, in patients with concomitant symptom cerebrovascular accidents (apoplectic ictus, etc.) are more prone to occur.]
* Patients with heart valve disease accompanied by pulmonary hypertension or fibrillary waves. Patients with heart valve disease with a history of acute bacterial endocardiosis [It has been reported that cardiovascular disorders such as thrombosis, etc. are liable to occur.]
* Patients with diabetes accompanied by vascular lesion (diabetic nephropathy, diabetic retinopathy, etc.) [It has been reported that cardiovascular disorders such as thrombosis, etc. are liable to occur.]
* Women with constitution of thrombosis [It has been reported that cardiovascular disorders including thrombosis, etc. are liable to occur.]
* Patients with antiphospholipid antibody syndrome [It has been reported that cardiovascular disorders including thrombosis, etc. are liable to occur.]
* Patient within 4 weeks before operation, within 2 weeks after operation, within 4 weeks of after delivery or at rest for a long-term period [Blood coagulation capacity is increased and the risk of occurrence of adverse reactions in the cardiovascular system may become high.]
* Patients with serious hepatic disorder [Since metabolic capacity is decreased, the burden on the liver increases, and the symptom may be aggravated.]
* Patients with hepatic tumor [The symptom may be aggravated.]
* Patients with lipid metabolism disorder [It has been reported that cardiovascular disorders including thrombosis, etc. are liable to occur. Since there is a possibility of lipid metabolism being affected, the symptom may be aggravated.]
* Patients with hypertension (excluding mild hypertension) [It has been reported that cardiovascular disorders including thrombosis, etc. are liable to occur. The symptom may be aggravated.]
* Patients with otosclerosis [The symptom may be aggravated.]
* Patients with a history of jaundice, persisting itching or gestational herpes during pregnancy [The symptom may be aggravated.]
* Pregnant or possibly pregnant women [Refer to the section "Use during Pregnancy, Delivery or Lactation".]
* Lactating women [Refer to the section "Use during Pregnancy, Delivery or Lactation".]
* Women before puberty [Early epiphysiodesis may occur.]

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be selected from clinical institutions where Marvelon® was adopted and delivered.
Sampling Method: Non-Probability Sample
Enrollment: 3838 (Actual)
Dates: Start 2005-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Number of participants who did not get pregnant during the study. | End of every 12 menstrual cycles up to 36 or at the termination of drug administration.